CLINICAL TRIAL: NCT05980273
Title: Effectiveness of Oral Health Education Programs Among School Children, Their Mothers and Teachers in Fayyum: Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yomna sayed khallaf, lecturer at faculty of dentistry Cairo university, Cairo University
Other Study IDs: health education -Oral Health
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Dental Caries
Keywords: oral health; Educational health program
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- school children, their mothers and teachers: educational session program
  Interventions: Behavioral: Educational sessions

INTERVENTIONS:
Behavioral: Educational sessions — session for oral health education

SUMMARY:
Cohort study to evaluate the effect of oral health educational program effect on oral health of school children, their mothers and teachers

DETAILED DESCRIPTION:
Scientific Background:

One of the most common disorders in the world is oral disease, which is mostly avoidable. In industrialized nations, dental caries affects 60-90% of schoolchildren and the majority of adults; it is becoming more common in developing nations and is particularly common in various Asian and Latin American nations .

Severe periodontitis affects 5-15% of the majority of people worldwide, and it is unmistakably linked to diabetes and weakened immune systems. Dental caries is common in India, where they affect 63.1% of 15-year-olds and up to 80.2% of individuals between the ages of 35 and 44, according to the National Oral Health Survey. Between the ages of 35 and 44, the prevalence of periodontal diseases increases to 89.6%, affecting 67.7% of 15-year-olds.

According to estimates, this chronic illness affects 60% to 90% of children who are of school age. This percentage fluctuates widely depending on the population, with the Middle East and other developing nations seeing higher rates of dental caries than wealthy nations do.

Any civilization that wants to give its citizens a fair standard of living should priorities preventing disease, disability, and pain. The most economical strategy and one that has the biggest influence on a community or population, whether it be a school, neighborhood, or country, is prevention on a community or population-based level. A planned action that delays the beginning of a disease among a population is known as an effective community preventative programs. There are many various ways to avoid dental diseases, but health education is the most economical one.

Numerous research on intermediate school students' awareness of oral health issues and use of preventative measures have been carried out. Rural Chinese pupils lacked understanding about fluoride use, gum disease, and dental caries. In Spain, 61.1% of 12-year-old children had at least one tooth that was decaying, filled, or missing, and they had little understanding of gingivitis. When knowledge in schoolchildren rose in the United Arab Emirates, practice also increased, demonstrating the connection between information and practice.

Only a few epidemiological studies of dental caries among Egyptians have been published, despite the significant frequency of dental caries in the community. Additionally, the majority of the information is in the form of grey literature and is not accessible through standard search engines. In 2014, the (WHO) and the Egyptian Ministry of Health conducted the most recent epidemiological assessment on the state of oral health in Egypt. Additionally, the majority of epidemiological research and only one ( focused on children.

To create and implement an effective children's oral health agenda and awareness programs for parents and school teachers that will enhance oral health, the prevalence of dental caries should be regularly monitored. Therefore, this study aimed to evaluate the prevalence of dental caries and periodontal diseases in mothers and children in fayoum, Egypt. Additionally, to evaluate the oral hygiene knowledge in mothers and children with enhancing prevention program.

ELIGIBILITY:
Inclusion Criteria:

* all students , their mothers & teachers will be included in this study

Exclusion Criteria:

* no exclusion criteria

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school children (7-14 years old) Their mothers children
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2023-10-09 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
oral health questionnaire | through one year
  Arabic version of a modified HU-DBI questionnaire

SECONDARY OUTCOMES:
decayed,missed,filled teeth / decayed , extracted , filled teeth | through one year
  decayed,missed,filled
Periodontal health/oral health status using BPE for mothers and teachers | through one year
  Code 0 Healthy Code 1 Bleeding on probing. No plaque retention factors or pockets greater than 3.5 mm Code 2 Presence of calculus or plaque retention factor. No pockets greater than 3.5 mm Code 3 Pockets of 3.5 to 5.5 mm Code 4 Pockets greater than 5.5 mm
  * Furcation involvement